CLINICAL TRIAL: NCT00117793
Title: Vacuum Suspension: Effects on Tissue Oxygenation, Activity and Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A3666
Record Dates: First submitted 2005-07-01; First posted 2005-07-08 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Amputation; Diabetes; Leg Injuries; Traumatic Amputations
Keywords: Amputee; Artificial limbs; Gait; Walking
MeSH Terms: conditions — Diabetes Mellitus; Leg Injuries; Amputation, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Current clinical practice
  Interventions: Device: Total Surface Bearing Suction Socket
- Arm 2 (Experimental): Novel socket system
  Interventions: Device: Vacuum assisted socket system

INTERVENTIONS:
Device: Total Surface Bearing Suction Socket — Current clinical practice
  Arms: Arm 1
Device: Vacuum assisted socket system — Novel socket system
  Arms: Arm 2

SUMMARY:
The fit of the residual limb within a prosthetic socket is a primary concern for many amputees. A poor fit can lead to skin irritation, tissue breakdown, and pain. Further, amputees with diabetes or vascular dysfunction often have difficulty maintaining healthy residual limb tissue; a condition that could be mitigated by the application of negative pressure (i.e., vacuum suspension). The aim of this research is to characterize the residual limb response to a vacuum suspension system and to measure prosthetic performance in comparison to a typical suction suspension system.

The proposed research plan involves two sets of human subject experiments: (1) prospective, randomized cross-over study to quantify performance of a vacuum suspension system as compared to a total surface bearing suction socket in terms of pistoning, maintaining limb volume, step counts, and subjective measures of fit and (2) measurement of transcutaneous oxygen tension as a function of vacuum pressure.

DETAILED DESCRIPTION:
A proper fitting prosthetic socket provides the amputee with a comfortable system allowing them to pursue many of their desired vocational and recreational goals. Unfortunately, many amputees live with an ill-fitting socket and can experience limb pistoning within the socket, which in turn may result in skin irritation, tissue breakdown, discomfort, and a reduction in activity. One of the key factors affecting fit is intraday residual limb volume changes. For an amputee with dysvascular conditions, the implications of a poor fitting socket are exacerbated by poor circulation, reduced healing potential and the compressive forces exerted by their prosthesis.

Vacuum suspension systems may have the potential to alleviate these conditions for healthy and dysvascular amputees. The purported benefits of vacuum suspension systems include, but are not limited to: improved suspension (reduction in the amount of pistoning), maintenance of limb volume throughout the day, and increased tissue oxygenation to the residual limb.

Our first objective is to characterize performance, as related to socket fit, of a vacuum suspension system using objective and subjective measures. We will do this by conducting a within-subject experiment to measure pistoning in three dimensions while walking, overall and regional changes in limb volume before and after a thirty-minute treadmill walk, mobility (step counts) and the perception of socket fit (questionnaire) as a function of prosthetic prescription (vacuum suspension system vs. total surface bearing suction socket).

Our second objective is to determine the effect of pressures within a prosthetic socket on residual limb transcutaneous oxygen tension (tcpO2) levels. We will conduct laboratory-based, in situ testing to determine how the transcutaneous oxygen tension levels, at six sites on the residual limb, respond to pressures simulating those within a vacuum suspension system and a total surface bearing suction socket.

The proposed research will allow us to understand how suspension systems influence prosthetic socket fit and residual limb tissue health and to formulate a knowledge base on two suspension systems providing prosthetists and clinicians the objective data to make better prescription decisions. In addition, the methods utilized in this study (e.g., a residual limb limb volume scanner and assessing dynamic pistoning) can be used to study current and novel suspension systems, liners, and prosthetic socket designs to provide a standard for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 and less than 70 years of age,
* Have a below knee amputation involving only one side,
* If the cause of amputation was for traumatic reasons and do not have diabetes or a vascular condition, the amputation must have occurred at least six months ago and the potential subject must have worn a prosthesis for at least four months,
* If the cause of amputation was for diabetes or vascular reasons, the potential subject must have been fit with a prosthesis and have worn it for at least one year,
* Wear the prosthesis for at least 6 hours a day,
* Able to walk without a cane, crutches, or a walker,
* Are moderately active enough to walk at a steady pace for at least 30 minutes.

Exclusion Criteria:

* Have pain in legs or any condition that interferes with walking.
* Have an ulcer on the residual limb,
* If potential subject had an amputation because of a tumor or an infection, no longer have an active tumor or undergoing treatment for a tumor,
* Have fallen within the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K. Klute, PhD, Principal Investigator — VA Puget Sound Health Care System, Seattle
Locations (1):
- VA Puget Sound Health Care System, Seattle, Seattle, Washington, United States

REFERENCES:
- [Derived] Klute GK, Berge JS, Biggs W, Pongnumkul S, Popovic Z, Curless B. Vacuum-assisted socket suspension compared with pin suspension for lower extremity amputees: effect on fit, activity, and limb volume. Arch Phys Med Rehabil. 2011 Oct;92(10):1570-5. doi: 10.1016/j.apmr.2011.05.019. PMID 21963124

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study was conducted at the VA Puget Sound Health Care System (Seattle VA hospital). Recruitment began on March 28, 2007. The study was closed to enrollment on March 30, 2012.
Pre-assignment Details: The prostheses used in this study were built and aligned by a certified and licensed prosthetist prior to beginning starting the protocol. 20 individuals gave informed consent but 3 withdrew prior to starting: 1 had contralateral knee surgery, 1 became a bi-lateral amputee, and 1 was withdrawn by the participant's physician.
Groups:
- Entire Study Population: This is a randomized cross-over study. Each participant wore both study prostheses: (1) a total surface bearing socket with a vacuum-assisted suspension system (VASS) and (2) a modified patellar tendon bearing socket with a pin lock suspension system (PIN).
  Subjects were randomized, provided with one of two study prostheses, and asked to wear it for three weeks. Data was then collected during laboratory visit one, and, following one more week of wearing the first study prosthesis, during laboratory visit two. Participants were then provided with the second study intervention and asked to wear it for three weeks. Data was then collected during laboratory visit three, and, following one more week of wearing the second study intervention, during laboratory visit four.
  Data was not collected on the order in which participants received each study intervention
Period: Overall Study
Arm/Group | Entire Study Population
Started | 17
Completed | 5
Not Completed | 12
Not completed — Withdrawal by Subject | 12

BASELINE CHARACTERISTICS:
Population: The sample population descriptors are based on the participants who completed the study protocol.
Groups:
- Entire Study Population: Includes participants randomized to receive PIN first and VASS first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Amputation etiology [Number; unit: Participants]
  Diabetic | 1
  Traumatic | 4
Years post-amputation [Mean (Standard Deviation); unit: Years] | 13 (15)
Weight [Mean (Standard Deviation); unit: kg] | 84 (11)
Height [Mean (Standard Deviation); unit: m] | 1.78 (0.11)

OUTCOME MEASURES:

1. Primary Outcome: Limb Volume
Time Frame: Measurements were taken after wearing the study prostheses for three weeks
Population: The number of participants for analysis is equal to the number of participants who completed the study protocol.
Measure: Mean (Standard Deviation); unit: liters
Groups:
- PIN Suspension: A modified patellar tendon bearing socket with a pin lock suspension system (PIN)
- VASS Suspension: A total surface bearing socket with a vacuum-assisted suspension system (VASS).
Arm/Group | PIN Suspension | VASS Suspension
Number analyzed (Participants) | 5 | 5
liters | 0.68 (.14) | 0.72 (.13)
Statistical Analysis 1: Comparison: PIN Suspension vs VASS Suspension; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — Statistical significance was set a-priori at p < 0.05; The effect of study limb on limb volume was analyzed using repeated measures one-way analyses of variance

2. Primary Outcome: Activity Level
Description: Total number of steps during a two week period ending in the fourth week for each study prosthesis (PIN and VASS).
Time Frame: Two weeks
Population: The number of participants for analysis is equal to the number of participants who completed the study protocol.
Measure: Mean (Standard Deviation); unit: steps (in thousands)
Arm/Group | PIN Suspension | VASS Suspension
Number analyzed (Participants) | 5 | 5
steps (in thousands) | 73 (18) | 38 (9)
Statistical Analysis 1: Comparison: PIN Suspension vs VASS Suspension; Test type: Superiority or Other; p = 0.0056, Mixed Models Analysis — Statistical significance was set a-priori at p < 0.05; The effect of study limb on activity level was analyzed using repeated measures one-way analyses of variance

3. Primary Outcome: Limb Pistoning
Description: Limb pistoning is the change in the resultant distance between the prosthetic-side knee joint marker triad and the residual limb thigh triad measured using a 12-camera motion analysis system while subjects weighted and un-weighted their prosthesis standing in place.
Time Frame: Measurements were taken after wearing the study prosthesis for three weeks
Population: The number of participants for analysis is equal to the number of participants who completed the study protocol.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PIN Suspension | VASS Suspension
Number analyzed (Participants) | 5 | 5
mm | 6 (4) | 1 (3)
Statistical Analysis 1: Comparison: PIN Suspension vs VASS Suspension; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis — Statistical significance was set a-priori at p < 0.05; The effect of study limb on limb pistoning was analyzed using repeated measures one-way analyses of variance

4. Secondary Outcome: Residual Limb Health (PEQ Scale)
Description: Qualitative differences between the study limbs were assessed using the Prosthesis Evaluation Questionnaire (PEQ). This standardized, self-report instrument is specific to persons with lower limb amputations and is used to evaluate prosthetic care with regard to prescription and prosthesis-related quality of life. The Residual Limb Health scale examines: sweat, smell, volume changes, rashes, ingrown hairs, and blisters. The scale is scored from 0 to 100 where 100 indicates the best outcome (i.e., most healthful).
Time Frame: Measurements were taken after wearing the study prosthesis for four weeks
Population: The number of participants for analysis is equal to the number of participants who completed the study protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PIN Suspension | VASS Suspension
Number analyzed (Participants) | 5 | 5
units on a scale | 90 (5) | 77 (20)

5. Secondary Outcome: Ambulation (PEQ Scale)
Description: Qualitative differences between the study limbs were assessed using the Prosthesis Evaluation Questionnaire (PEQ). This standardized, self-report instrument is specific to persons with lower limb amputations and is used to evaluate prosthetic care with regard to prescription and prosthesis-related quality of life. The Ambulation scale queries the ability to walk in general, in close spaces, on stairs and ramps, in urban environments, and on slippery surfaces. The scale is scored from 0 to 100 where 100 indicates the best outcome (i.e., easiest to walk on).
Time Frame: Measurements were taken after wearing the study prosthesis for four weeks
Population: The number of participants for analysis is equal to the number of participants who completed the study protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PIN Suspension | VASS Suspension
Number analyzed (Participants) | 5 | 5
units on a scale | 95 (6) | 67 (22)

6. Secondary Outcome: Frustration (PEQ Scale)
Description: Qualitative differences between the study limbs were assessed using the Prosthesis Evaluation Questionnaire (PEQ). This standardized, self-report instrument is specific to persons with lower limb amputations and is used to evaluate prosthetic care with regard to prescription and prosthesis-related quality of life. Frustration was assessed by frequency of occurrence and rating. The scale is scored from 0 to 100 where 100 indicates the best outcome (i.e., least frustrating).
Time Frame: Measurements were taken after wearing the study prosthesis for four weeks
Population: The number of participants for analysis is equal to the number of participants who completed the study protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PIN Suspension | VASS Suspension
Number analyzed (Participants) | 5 | 5
units on a scale | 91 (11) | 43 (29)

ADVERSE EVENTS:
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population (N=17)
Prosthesis failure (Injury, poisoning and procedural complications) | 1 (1) — Socket fracture during routine activity preventing further use. Participant was wearing VASS at time of failure.

LIMITATIONS AND CAVEATS:
The small number of participants who completed the protocol precluded a statistical analysis on the secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes